CLINICAL TRIAL: NCT05432674
Title: Digital Fall Prevention Feasibility Study
Brief Title: Digital Fall Prevention Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Best Buy Health, Inc (Unknown)
Responsible Party: Principal Investigator, Nancy Latham, Clinical Research Director, Research Division of Men's Health, Aging and Metabolism, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022P000630
Record Dates: First submitted 2022-06-17; First posted 2022-06-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Fall
Keywords: exercise; fall prevention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Fall Prevention (Experimental): Subjects will participate in Digital Fall Prevention intervention for 12 weeks
  Interventions: Combination Product: Digital Fall Prevention

INTERVENTIONS:
Combination Product: Digital Fall Prevention — Exercises delivered through a tablet and remote motivational calls

SUMMARY:
The Digital Fall Prevention Study is a single-group unblinded study to explore the feasibility and acceptability of a 3-month fall prevention exercise program delivered digitally via a tablet interface. Evidence-based exercise programs and motivational techniques will be used along with new wearable technology to predict fall risk.

DETAILED DESCRIPTION:
The goal of this study is to demonstrate the feasibility and acceptability of a digital fall prevention exercise program and to explore whether there is benefit from participating in such programs. This study will include 30 older adults who are at higher risk of falling or have a fear of falling and living at home. All participants will receive the intervention. All participants will be assessed pre- and post-intervention on measures of sensor-based fall risk, sensor-based frailty, falls self-efficacy, technology readiness, feasibility and acceptability, utilization and participation, frailty, grip strength, depression, anxiety, and physical activity (both self-report and using wearable sensors).

The overall hypothesis is that a prototype system consisting of wearable sensors and a tablet will be feasible and acceptable in a population of older adults with increased risk for falls and fall-related injuries or with a fear of falling.

Aim 1: To determine the feasibility and acceptability of a self-guided, digitally delivered, in-home exercise program for older adults with elevated fall risk.

* Hypothesis 1a): The technology (wearable sensor and tablet) and digitally delivered fall prevention exercises will be feasible and acceptable to older people at risk for falls.
* Hypothesis 1b): The technology (wearable sensor and tablet) and digitally delivered fall prevention exercise program will reduce a user's concern of falling

Aim 2: To determine the clinical effects of implementing a fall prevention intervention program via the remote platform.

• Hypothesis 2): Participants who adhere to the program, completing at least 70% of the video exercise sessions, will see a pre- to post-intervention reduction in quantitative measures of fall risk.

Exploratory Aim 1: Investigate differences in frailty, cognitive status, physical function, mental health status and technology readiness between participants who successfully adhere to the study program versus those that do not.

The study will take place in two settings. The first setting is at the Men's Health, Aging, and Metabolism research division at Brigham and Women's Hospital, including the Laboratory of Exercise Physiology and Physical Performance (LEPPP) at 221 Longwood Ave, Boston, MA 02115. The second will be in the homes of older adults within the general community who meet the inclusion criteria.

Intervention

Participants who enroll in the study will receive a wearable device, a tablet, a tablet stand, and ankle weights for home use, along with instructions and charging accessories. Participants will participate in a 3-month moderate-intensity exercise intervention, which will be supported by a LEPPP study staff member trained and certified in the intervention and delivered remotely through the tablet. The program is designed to gradually progress in intensity and exercise duration over a 12-week period. The exercise intervention parameters will be tailored to individual ability and progressed by the study interventionist based on feedback from participants, motivational coaching calls, and post-exercise surveys.

ELIGIBILITY:
Inclusion Criteria:

* Male and females who are 65 years or older
* Short Physical Performance Battery (SPPB)7 ≥ 5
* the Montreal Cognitive Assessment (MoCA)8 > 17
* Increased risk for falls based on a self-reported answer of yes to one or more of these questions:

  * Have you fallen and hurt yourself in the past year?
  * Have you fallen two or more times in the past year?
  * Are you afraid that you might fall because of balance or walking problems?
* Access to Wi-Fi in their home (or willingness to use cellular service if provided)

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* MI, acute coronary syndrome, revascularization surgery, or stroke in the last 6 months
* Chest pain or untreated/uncontrolled CVD
* Hip/knee fracture/replacement or spinal surgery in past 6 months
* Pulmonary decompensation that would prevent participation in the exercise program
* Planned orthopedic surgery that would limit participation in the study
* Planned to be away from tablet access for > 7 days during the length of the study
* Unable to attend in-person pre- or post-study clinic visit
* Enrolled in a formal exercise program and/or physical therapy that takes place 3 or more times per week
* Vision or hearing impairments that would make it difficult to participate in the intervention
* Non-English speaking or other language limitations that would make it difficult to participate in the intervention
* Reside in a nursing home
* Unable to walk independently (with or without a walking aid)
* Not appropriate for study based on clinician exam or discretion (clinician will specify reason)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Acceptability and adherence to exercise program | over the 12 weeks of the intervention
  Percentage of scheduled exercise sessions complete (70% of sessions completed = acceptable adherence)
Feasibility of Intervention Measure (FIM) | at final (12-week) assessment
  a self-report measure of the intervention feasibility, score range is 1-5, higher score = greater feasibility
Acceptability of Intervention Measure (AIM) | at final (12-week) assessment
  a self-report measure of acceptability of the intervention, score range is 1-5, higher score = greater acceptability
Fall Efficacy Scale - International (FES-I) | change from baseline to 12-weeks
  fear of falling measure, score range from 16-64, higher score=less fear of falling
Intervention Appropriateness Measure (IAM) | at final (12-week) assessment
  a self-report measure of the intervention appropriateness, score range is 1-5, higher score = greater appropriateness

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | change from baseline to 12-weeks
  cognitive status assessment, score range 0-30, higher score=better cognition
Digit Symbol Substitution Test | change from baseline to 12-weeks
  cognitive assessment
Fried Frailty Index (FFI) | change from baseline to 12-weeks
  measure of frailty in older people, index range from 1-5, higher score=increased frailty
Grip Strength of dominant hand | change from baseline to 12-weeks
  maximal isometric contraction of hand measured using a Jamar Handheld Dynamometer in kilograms
  Strength (force) will be measured in kilograms.
Physical Activity Scale for the Elderly (PASE) | change from baseline to 12-weeks
  self-report physical activity scale, score range 0 to 400, higher score=more activity
Sensor based fall risk assessment | change from baseline to 12-weeks
  fall risk assessed using a sensor and computer based program
Sensor based frailty assessment | change from baseline to 12-weeks
  frailty assessed using a sensor and computer based program
Short Physical Performance Battery (SPPB) | change from baseline to 12-weeks
  physical performance mobility test
Technology Acceptance Model (TAM) | at final (12-week) assessment
  a self-report measure of the acceptance of the technology used in the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kieran F Reid, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No